CLINICAL TRIAL: NCT00295633
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled, Phase III Trial to Evaluate the Efficacy and Safety of Saxagliptin (BMS477118) in Combination With Thiazolidinedione Therapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Thiazolidinedione Therapy Alone
Brief Title: A Study Assessing Saxagliptin Treatment in Type 2 Diabetic Subjects Who Are Not Controlled With TZD Therapy Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV181-013
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Results first posted 2009-09-25 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Pioglitazone; Rosiglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Saxagliptin plus open-label TZD (A) (Experimental): Saxagliptin PLUS pioglitazone OR rosiglitazone
  PLUS open-label metformin (as needed as rescue medication)
  Interventions: Drug: Saxagliptin; Drug: pioglitazone; Drug: rosiglitazone; Drug: metformin
- Saxagliptin plus open-label TZD (B) (Experimental): Saxagliptin PLUS pioglitazone OR rosiglitazone
  PLUS open-label metformin (as needed as rescue medication)
  Interventions: Drug: Saxagliptin; Drug: pioglitazone; Drug: rosiglitazone; Drug: metformin
- Placebo plus open-label TZD (C) (Placebo Comparator): Placebo PLUS pioglitazone OR rosiglitazone
  PLUS open-label metformin (as needed as rescue medication)
  Interventions: Drug: Placebo; Drug: pioglitazone; Drug: rosiglitazone; Drug: metformin

INTERVENTIONS:
Drug: Saxagliptin — Tablets, Oral, 2.5 mg, Once daily (6 months ST, 12 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin plus open-label TZD (A)
Drug: Saxagliptin — Tablets, Oral, 5 mg, once daily (6 months ST, 12 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin plus open-label TZD (B)
Drug: Placebo — Tablets, Oral, 0 mg, Once daily (6 months ST, 12 months LT)
  Arms: Placebo plus open-label TZD (C)
Drug: pioglitazone — Tablets, Oral, 30 mg or 45 mg, once daily (6 months ST, 12 months LT)
Drug: rosiglitazone — Tablets, Oral, 4 mg, once daily or 8 mg, either as once or twice daily (6 months ST, 12 months LT)
Drug: metformin — Tablets, Oral, 500-2500 mg, as needed (12 months LT)

SUMMARY:
The purpose of this clinical research study is to learn whether Saxagliptin added to thiazolidinedione (TZD) therapy is more effective than TZD alone as a treatment for Type 2 diabetic subjects who are not sufficiently controlled with TZD alone

DETAILED DESCRIPTION:
All subjects will participate in a lead-in period, and qualifying subjects will continue into a short-term randomized treatment period. Subjects who complete the short-term period will be eligible to enter the long term extension period. Also, subjects in the short-term period who have an elevated blood sugar that requires additional medication for blood sugar control will be eligible to enter the long-term treatment extension period where they will receive metformin (defined as rescue medication) added onto their blinded study medication

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetics currently receiving a stable dose of TZD monotherapy (pioglitazone 30mg or 45mg, or rosiglitazone 4mg or 8mg) for at least 12 weeks prior to screening.
* Hemoglobin A1c (HbA1c) > = 7.0% and < = 10.5%
* Body mass index < = 45kg/m2
* Fasting C-peptide > = 1 ng/mL

Exclusion Criteria:

* Symptomatic poorly controlled diabetes
* Recent cardiac or cerebrovascular event
* Serum creatinine > = 2.0 mg/dL

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (126):
- United States (79):
  - Winston Technology, Inc., Haleyville, Alabama
  - Sunbelt Research Group, Llc, Mobile, Alabama
  - Iicr, Inc., Ozark, Alabama
  - Clinical Research Advantage, Inc, Mesa, Arizona
  - Nea Clinic, Jonesboro, Arkansas
  - Little Rock Family Practice Clinic, Little Rock, Arkansas
  - Impact Clinical Trials, Beverly Hills, California
  - Lovelace Scientific Resources, Inc., Beverly Hills, California
  - Medical Group Of Encino, Encino, California
  - Marin Endocrine Care And Research, Inc., Greenbrae, California
  - Del Rosario Medical Clinic, Inc., Huntington Park, California
  - Loma Linda Va Healthcare Systems, Loma Linda, California
  - Peak Health Medical Group, Los Angeles, California
  - Richard Cherlin, Md, Los Gatos, California
  - Mission Internal Medical Group, Mission Viejo, California
  - Desert Medical Advances, Palm Desert, California
  - Denver Internal Medicine Group, Denver, Colorado
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Phoenix Internal Medicine Associates, Llc, Waterbury, Connecticut
  - Central Florida Clinical Trials, Inc., Altamonte Springs, Florida
  - Southern Family Healthcare, Pa, Chipley, Florida
  - Doctors Medical Center Of Walton County, DeFuniak Springs, Florida
  - Horizon Institute For Clinical Research, Hollywood, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Panhandle Family Care Associates, Marianna, Florida
  - Nextphase Clinical Trials, Inc, Miami, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - Heart & Vascular Center Research, Inc., Sarasota, Florida
  - Alan B. Miller, Md, Dunwoody, Georgia
  - Marietta Clinical Research, Inc., Marietta, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - D. Thomas Rogers, Md, Facs, Kahului, Hawaii
  - Southeast Idaho Family Practice, Idaho Falls, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Physicians Research Group, Indianapolis, Indiana
  - Northwest Indiana Center For Clinical Research, Valparaiso, Indiana
  - Lipid Research Clinic, Iowa City, Iowa
  - Professional Research Network Of Kansas, Wichita, Kansas
  - Mouhaffel, Assad H., West Monroe, Louisiana
  - Promed Physicians Family Practice, Portage, Michigan
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Radiant Research Las Vegas, Las Vegas, Nevada
  - Nevada Alliance Against Diabetes, North Las Vegas, Nevada
  - Office Of Ammar Bazerbashi, Md, Holmdel, New Jersey
  - Urgentmed, P.C., South Bound Brook, New Jersey
  - Medical Research Associates Of Charlotte, Inc., Charlotte, North Carolina
  - Carolina Pharmaceutical Research, Statesville, North Carolina
  - Community Health Care, Canal Fulton, Ohio
  - Clinical Research Limited, Canton, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Providence Health Partners - Center For Clinical Research, Dayton, Ohio
  - Holzer Clinic, Gallipolis, Ohio
  - Wells Institute For Health Awareness, Kettering, Ohio
  - David Witkin, Md, Eugene, Oregon
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Family Medical Associates, Levittown, Pennsylvania
  - Banksville Medical Pc, Pittsburgh, Pennsylvania
  - Three Rivers Medical Associates, Pa, Columbia, South Carolina
  - Radiant Research, Greer, Greer, South Carolina
  - Upstate Pharmaceutical Research, Simpsonville, South Carolina
  - East Tennessee Medical Group, Alcoa, Tennessee
  - Healthstar Physicians, Morristown, Tennessee
  - Hayes Endocrine And Diabetes Center, Nashville, Tennessee
  - Capital Medical Clinic, Llp, Austin, Texas
  - Texas Diabetes And Endocrinology, P.A., Austin, Texas
  - Radiant Research-Austin, Austin, Texas
  - Priscilla Hollander, Md, Phd, Dallas, Texas
  - The Medical Group Of Texas, Fort Worth, Texas
  - Mobley Research Center, Houston, Texas
  - Family Physician, Pa, Houston, Texas
  - Mapleridge Medical Center, Houston, Texas
  - Diabetes Center Of The Southwest, Midland, Texas
  - Pearland Primary Care Associates, Llp, Pearland, Texas
  - Med-Cure, Rosenberg, Texas
  - Radiant Research San Antonio, San Antonio, Texas
  - S.A.M. Clinical Research Center, San Antonio, Texas
  - Collom And Carney Clinic, Texarkana, Texas
  - National Clinical Research, Inc., Richmond, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
- Argentina (10):
  - Local Institution, Belgrano, Buenos Aires
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Chacabuco, Buenos Aires
  - Local Institution, Ciudad Auton., Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Morón, Buenos Aires
  - Local Institution, Mendoza, Mendoza Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Lanus Este, Tucumán Province
  - Local Institution, Buenos Aires
- Canada (7):
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Sarnia, Ontario
  - Local Institution, St. Catharines, Ontario
  - Local Institution, Saint-Léonard, Quebec
  - Local Institution, Ste-Foy, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- India (10):
  - Local Institution, Bangalore
  - Local Institution, Chennai
  - Local Institution, Hariyāna
  - Local Institution, Hyderabad
  - Local Institution, Indore
  - Local Institution, Maharashtra
  - Local Institution, Mangalore
  - Local Institution, Mumbai
  - Local Institution, Pune
  - Local Institution, Vellore
- Mexico (6):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Chichuahua, Chihuahua
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Angeles Del Pedregal, Mexico City
  - Local Institution, Michoacan, Morelos
  - Local Institution, Monterrey, Nuevo León
- Peru (6):
  - Local Institution, La Victoria, Lima region
  - Local Institution, Lima Cercado, Lima region
  - Local Institution, Miraflores, Lima region
  - Local Institution, San Isidro, Lima region
  - Local Institution, San Martín de Porres, Lima region
  - Local Institution, Santiago de Surco, Lima region
- Philippines (4):
  - Local Institution, Cebu City
  - Local Institution, Iloilo City
  - Local Institution, Las Piñas
  - Local Institution, Pasig
- Puerto Rico (4):
  - Local Institution, Carolina
  - Local Institution, Ponce
  - Local Institution, Rio Piedras
  - Local Institution, San Juan

REFERENCES:
- [Background] Hollander P, Li J, Allen E, Chen R; CV181-013 Investigators. Saxagliptin added to a thiazolidinedione improves glycemic control in patients with type 2 diabetes and inadequate control on thiazolidinedione alone. J Clin Endocrinol Metab. 2009 Dec;94(12):4810-9. doi: 10.1210/jc.2009-0550. Epub 2009 Oct 28. PMID 19864452
- [Derived] Perl S, Cook W, Wei C, Iqbal N, Hirshberg B. Saxagliptin Efficacy and Safety in Patients With Type 2 Diabetes and Moderate Renal Impairment. Diabetes Ther. 2016 Sep;7(3):527-35. doi: 10.1007/s13300-016-0184-9. Epub 2016 Jul 11. PMID 27402391
- [Derived] Bonora E, Bryzinski B, Hirshberg B, Cook W. A post hoc analysis of saxagliptin efficacy and safety in patients with type 2 diabetes stratified by UKPDS 10-year cardiovascular risk score. Nutr Metab Cardiovasc Dis. 2016 May;26(5):374-9. doi: 10.1016/j.numecd.2015.11.004. Epub 2015 Dec 1. PMID 27033025
- [Derived] Karyekar CS, Frederich R, Ravichandran S. Clinically relevant reductions in HbA1c without hypoglycaemia: results across four studies of saxagliptin. Int J Clin Pract. 2013 Aug;67(8):759-67. doi: 10.1111/ijcp.12212. Epub 2013 Jun 24. PMID 23795975
- [Derived] Karyekar C, Donovan M, Allen E, Fleming D, Ravichandran S, Chen R. Efficacy and safety of saxagliptin combination therapy in US patients with type 2 diabetes. Postgrad Med. 2011 Jul;123(4):63-70. doi: 10.3810/pgm.2011.07.2305. PMID 21680990
- [Derived] Hollander PL, Li J, Frederich R, Allen E, Chen R; CV181013 Investigators. Safety and efficacy of saxagliptin added to thiazolidinedione over 76 weeks in patients with type 2 diabetes mellitus. Diab Vasc Dis Res. 2011 Apr;8(2):125-35. doi: 10.1177/1479164111404575. PMID 21562064

RESULTS

PARTICIPANT FLOW:
Groups:
- Saxagliptin 2.5 mg Plus Open-label Thiazolidinedione (TZD): The Saxagliptin 2.5 mg + Open-Label TZD group includes data from subjects randomized to receive coadministration of blinded Saxagliptin 2.5 mg plus open-label pioglitazone 30 mg or 45 mg once daily (QD), or open label rosiglitazone 4 mg QD, or 8 mg, either QD or in 2 divided doses of 4 mg.
- Saxagliptin 5 mg Plus Open-label TZD: The Saxagliptin 5 mg + Open-Label TZD group includes data from subjects randomized to receive coadministration of blinded Saxagliptin 5 mg plus pioglitazone 30 mg or 45 mg once daily (QD), or rosiglitazone 4 mg QD, or 8 mg, either QD or in 2 divided doses of 4 mg.
- Placebo Plus Open-label TZD: The placebo + open-label TZD group includes data from subjects randomized to receive coadministration of blinded placebo plus pioglitazone 30 mg or 45 mg once daily (QD), or rosiglitazone 4 mg QD, or 8 mg, either QD or in 2 divided doses of 4 mg.
Period: Overall Study
Arm/Group | Saxagliptin 2.5 mg Plus Open-label Thiazolidinedione (TZD) | Saxagliptin 5 mg Plus Open-label TZD | Placebo Plus Open-label TZD
Started | 195 | 186 | 184
Completed Study Without Being Rescued | 88 | 82 | 51
Completed | 133 | 119 | 108
Not Completed | 62 | 67 | 76
Not completed — Lack of Efficacy | 19 | 7 | 16
Not completed — Withdrawal of consent by subject | 16 | 16 | 26
Not completed — Adverse Event | 9 | 17 | 9
Not completed — Lost to Follow-up | 6 | 11 | 7
Not completed — Physician Decision | 9 | 10 | 8
Not completed — Poor/Noncompliance | 2 | 2 | 6
Not completed — Subject No Longer Meets Study Criteria | 0 | 3 | 3
Not completed — Death | 1 | 1 | 0
Not completed — Administrative reason by sponsor | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Saxagliptin 2.5 mg Plus Open-label TZD: The Saxagliptin 2.5 mg + Open-Label TZD group includes data from subjects randomized to receive coadministration of blinded Saxagliptin 2.5 mg plus open-label pioglitazone 30 mg or 45 mg once daily (QD), or open label rosiglitazone 4 mg QD, or 8 mg, either QD or in 2 divided doses of 4 mg.
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 2.5 mg Plus Open-label TZD | Saxagliptin 5 mg Plus Open-label TZD | Placebo Plus Open-label TZD | Total
Number analyzed (Participants) | 195 | 186 | 184 | 565
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.85 (9.73) | 53.22 (10.56) | 54.01 (10.08) | 54.04 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 97 | 99 | 285
  Male | 106 | 89 | 85 | 280

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (A1C) at Week 24
Description: Mean change from baseline in A1C at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis of change from baseline to Week 24 Last Observation Carried Forward (LOCF), participants must have had a baseline and at least 1 post-baseline measurement. If participant received rescue medication, measurement must have been taken before rescue.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Saxagliptin 2.5 mg Plus Open-label TZD | Saxagliptin 5 mg Plus Open-label TZD | Placebo Plus Open-label TZD
Number analyzed (Participants) | 192 | 183 | 180
percent
  Baseline Mean | 8.25 (0.080) | 8.35 (0.080) | 8.19 (0.080)
  Week 24 Mean | 7.59 (0.098) | 7.39 (0.086) | 7.91 (0.100)
  Adjusted Mean Change from Baseline | -0.66 (0.074) | -0.94 (0.075) | -0.30 (0.076)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Mean change from baseline in FPG at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis of change from baseline to Week 24 LOCF, participants must have had a baseline and at least 1 post-baseline measurement. If a participant received rescue medication, then that measurement must have been taken before rescue.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg Plus Open-label TZD | Saxagliptin 5 mg Plus Open-label TZD | Placebo Plus Open-label TZD
Number analyzed (Participants) | 193 | 185 | 181
mg/dL
  Baseline Mean | 163.0 (3.54) | 159.5 (3.34) | 162.4 (3.43)
  Week 24 Mean | 148.2 (3.36) | 143.0 (3.20) | 159.3 (4.29)
  Adjusted Mean Change from Baseline | -14.3 (2.87) | -17.3 (2.94) | -2.8 (2.97)

3. Secondary Outcome: Percentage of Participants Achieving A1c <7% at Week 24
Description: Percentage of participants achieving A1C < 7%, the American Diabetic Association's defined goal for glycemia, at each dose of saxagliptin plus TZD versus placebo plus TZD at Week 24.
Time Frame: Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in the Week 24 LOCF analysis, subjects must have had at least 1 post-baseline measurement. If a participant received rescue medication, then that measurement must have been taken before rescue.
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 2.5 mg Plus Open-label TZD | Saxagliptin 5 mg Plus Open-label TZD | Placebo Plus Open-label TZD
Number analyzed (Participants) | 192 | 184 | 180
Percentage of participants | 42.2 | 41.8 | 25.6

4. Secondary Outcome: Changes From Baseline in Postprandial Glucose (PPG) Area Under the Curve (AUC) Response to an Oral Glucose Tolerance Test (OGTT) at Week 24
Description: Mean change from baseline for 0 to 180 minutes PPG AUC achieved at each dose of saxagliptin plus TZD versus placebo plus TZD at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Saxagliptin 2.5 mg Plus Open-label TZD | Saxagliptin 5 mg Plus Open-label TZD | Placebo Plus Open-label TZD
Number analyzed (Participants) | 151 | 131 | 123
mg*min/dL
  Baseline Mean | 48301 (968.5) | 47866 (1048.9) | 47256 (1057.4)
  Week 24 Mean | 40255 (919.7) | 38587 (991.3) | 44819 (1023.4)
  Adjusted Mean Change from Baseline | -7849 (740.6) | -9269 (794.9) | -2690 (820.6)

ADVERSE EVENTS:
Arm/Group | PLA + TZD | SAXA 2.5MG + TZD | SAXA 5MG + TZD
Serious Adverse Events (participants affected / at risk) | 20/184 | 19/195 | 18/186
Other Adverse Events (participants affected / at risk) | 109/184 | 107/195 | 109/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLA + TZD (N=184) | SAXA 2.5MG + TZD (N=195) | SAXA 5MG + TZD (N=186)
CATARACT (Eye disorders) | 0 | 1 | 0
BLOOD PRESSURE INCREASED (Investigations) | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 3 | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 1
ALCOHOL ABUSE (Psychiatric disorders) | 0 | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 2 | 0
CEREBRAL HAEMATOMA (Nervous system disorders) | 0 | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1 | 0
CEREBELLAR HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 1 | 0
ANAL FISTULA (Gastrointestinal disorders) | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 0 | 1
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0
ORCHITIS (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0 | 1
ANAL ABSCESS (Infections and infestations) | 0 | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 2 | 1
MENINGITIS ASEPTIC (Infections and infestations) | 1 | 0 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0 | 0
RENAL CYST (Renal and urinary disorders) | 0 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0 | 1
CALCULUS BLADDER (Renal and urinary disorders) | 0 | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 | 0 | 1
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 | 0 | 1
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 1
BACK INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PYREXIA (General disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 1 | 1 | 1
SUDDEN DEATH (General disorders) | 0 | 0 | 1
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PLA + TZD (N=184) | SAXA 2.5MG + TZD (N=195) | SAXA 5MG + TZD (N=186)
HYPERTENSION (Vascular disorders) | 12 | 15 | 11
HEADACHE (Nervous system disorders) | 12 | 15 | 15
DIZZINESS (Nervous system disorders) | 14 | 10 | 7
DIARRHOEA (Gastrointestinal disorders) | 13 | 8 | 10
BRONCHITIS (Infections and infestations) | 9 | 11 | 7
NASOPHARYNGITIS (Infections and infestations) | 15 | 9 | 15
URINARY TRACT INFECTION (Infections and infestations) | 17 | 23 | 20
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 19 | 25 | 24
ANAEMIA (Blood and lymphatic system disorders) | 3 | 3 | 11
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 12 | 12
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 13 | 22 | 10
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 6 | 10 | 12
COUGH (Respiratory, thoracic and mediastinal disorders) | 13 | 9 | 5
PYREXIA (General disorders) | 8 | 6 | 11
OEDEMA PERIPHERAL (General disorders) | 19 | 9 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.